CLINICAL TRIAL: NCT04796584
Title: Efficacy of COVID 19 SARS-CoV-2 mRNA Vaccination in Patients With Multiple Sclerosis Treated With Immune Modulating Medication (SARSmRNA_MS)
Brief Title: Efficacy of COVID-19 Vaccination in Patients With Multiple Sclerosis Treated With Immune Modulating Medication
Status: Terminated | Type: Observational
Why Stopped: Enrollment paused for greater than 6 months, data would not be relevant as enrollment took longer than expected.
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Other Study IDs: SARSmRNA_MS
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: mRNA-based SARS-CoV-2 vaccination
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples will be analyzed for the presence and titer of neutralizing antibodies to the SARSCoV-2 virus. Isolated peripheral blood lymphocytes will be used for analyses of T cell responses to SARS-CoV-2 spike peptides.
  The unused portion of the samples will be stored for future deep cytokine and genomic analyses if funding becomes available to perform these latter studies. Data and samples will be stored indefinitely. It is possible that disease specific genetic testing, as it relates to the Donor's diagnosis of autoimmunity and their immune response to the vaccine and/or their autologous tissue, may be done on samples. Other testing may be done as technology and scientific knowledge about the immune response to vaccines and autoimmunity advances
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MS subjects who are being treated with ocrelizumab: Ocrelizumab's immunomodulating mechanisms of action is B-cell lytic. Each consenting subject will provide approximately 30 mL of whole blood via venipuncture before and 45, 90 and 180 days after the first vaccine injection and 28-42 days after the booster vaccination (if applicable).
  Interventions: Other: Analysis of cell-mediated and antibody-mediated immunity to SARS-CoV-2 virus
- MS subjects who are being treated with fingolimod: Fingolimod's immunomodulating mechanisms of action is to prevent mobilization of B and T cells from peripheral lymphoid organs. Each consenting subject will provide approximately 30 mL of whole blood via venipuncture before and 45, 90 and 180 days after the first vaccine injection and 28-42 days after the booster vaccination (if applicable).
  Interventions: Other: Analysis of cell-mediated and antibody-mediated immunity to SARS-CoV-2 virus
- MS subjects who are being treated with natalizumab: Natalizumab's immunomodulating mechanisms of action is to block transmigration of monocytes, and lymphocytes into the central nervous system. Each consenting subject will provide approximately 30 mL of whole blood via venipuncture before and 45, 90 and 180 days after the first vaccine injection and 28-42 days after the booster vaccination (if applicable).
  Interventions: Other: Analysis of cell-mediated and antibody-mediated immunity to SARS-CoV-2 virus
- MS subjects who are being treated with dimethyl fumarate/diroximel fumarate: Dimethyl Fumarate's immunomodulating mechanisms of action is to reduce inflammation-induced oxidative stress. Each consenting subject will provide approximately 30 mL of whole blood via venipuncture before and 45, 90 and 180 days after the first vaccine injection and 28-42 days after the booster vaccination (if applicable).
  Interventions: Other: Analysis of cell-mediated and antibody-mediated immunity to SARS-CoV-2 virus

INTERVENTIONS:
Other: Analysis of cell-mediated and antibody-mediated immunity to SARS-CoV-2 virus — mRNA vaccination for SARS-CoV-2 is not provided by the study

SUMMARY:
The primary objective is to determine whether the use of immunomodulating medications have an impact on the ability to mount and sustain an immune response to SARS-CoV-2 spike protein following mRNA vaccination in patients with MS when compared to healthy controls not receiving immunomodulating medications.

We hypothesize that the use of immunomodulators in MS patients may eliminate or reduce the level of protective immune response, and/or shorten the duration of the protective response.

DETAILED DESCRIPTION:
Analysis of cell-mediated and antibody-mediated immunity to the COVID-19, SARS-CoV-2 virus following treatment with mRNA vaccine, in patients with multiple sclerosis (MS) who are treated with immune modulating medication. Each consenting subject will provide approximately 30 mL of whole blood via venipuncture before their first vaccine injection (those who meet inclusion 3a only), 45 (those who meet inclusion 3a or 3b), 90 and 180 days after the first vaccine injection (those who meet inclusion 3a, 3b, or 3c). If they receive a booster vaccine injection, they will also be asked to provide 30 mL of whole blood 28-42 days after the booster injection date. These samples, obtained at Providence St. Vincent Medical Center, will be transferred to the Laboratory of Molecular and Tumor Immunology at the Earle A. Chiles Cancer Research Institute, where the blood will be processed and cryopreserved. Serum samples will be analyzed for the presence and titer of neutralizing antibodies to the SARS-CoV-2 virus. Isolated peripheral blood lymphocytes will be used for analyses of T cell responses to SARS-CoV-2 spike peptides. Responses will be compared to the immune responses of 10 subjects who have been enrolled in the CORVax spike plasmid DNA vaccine study and are subsequently referred to in this protocol as "healthy controls." The unused portion of the samples will be stored for future deep cytokine and genomic analyses if funding becomes available to perform these latter studies.

This study will include 4 cohorts, each will enroll 10 subjects who are being treated with an immunomodulating therapy for MS. The 4 immunomodulating medications selected, because each differs in their mechanisms of action, include ocrelizumab (B-cell lytic), fingolimod (prevents mobilization of B and T cells from peripheral lymphoid organs), natalizumab (blocks transmigration of monocytes, and lymphocytes into the central nervous system), and dimethyl fumarate/diroximel fumarate (reduces inflammation-induce oxidative stress).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose, benefits, and risks of the study; willing and able to adhere to the study requirements; able to provide informed consent in English
2. Male or female, between the ages of 18 and 65 years inclusive at time of consent
3. Meet one of the following:

   1. Plan to receive one of the FDA approved mRNA-based COVID SARS-CoV-2 vaccinations within 30 days of the screening visit
   2. Have received one of the FDA approved mRNA-based COVID SARS-CoV-2 vaccinations, their first vaccine injection having occurred 45±7 days prior to the screening visit
   3. Have received one of the FDA approved mRNA-based COVID SARS-CoV-2 vaccinations, their first vaccine injection having occurred 90±7 days prior to the screening visit
4. Meet the criteria of one of the four groups at the time of consent:

Group 1: Diagnosed with multiple sclerosis and currently being treated with a stable dose of ocrelizumab, for 6 months or longer Group 2: Diagnosed with multiple sclerosis and currently being treated with a stable dose of fingolimod, for 6 months or longer Group 3: Diagnosed with multiple sclerosis and currently being treated with a stable dose of natalizumab, for 6 months or longer Group 4: Diagnosed with multiple sclerosis and currently being treated with a stable dose of dimethyl fumarate or diroximel fumarate, for 6 months or longer

Exclusion Criteria:

1. Subjects who have a BMI of >35.0 will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There is no available information on whether patients being treated with immunomodulating agents will mount a response to SARS-CoV-2 vaccination comparable to that observed in the general population. Volunteers will be recruited from the MS patient population cared for at the Providence MS Center. Patients will be identified by review of electronic medical records. Patients who appear to meet the eligibility criteria will be contacted by an investigator and/or a delegated research staff member.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Titer of antibody against SARS-CoV-2 spike protein | Day 45 following initial vaccination
  Serum Sample
Quantity of IFN-g secreted in response to stimulation with SARS-CoV-2 spike protein | Day 45 following initial vaccination
  Serum Sample
Quantity of TNF-a secreted in response to stimulation with SARS-CoV-2 spike protein | Day 45 following initial vaccination
  Serum Sample

SECONDARY OUTCOMES:
Titer of antibody against SARS-CoV-2 spike protein | Day 90 following initial vaccination
  Serum Sample
Quantity of IFN-g secreted in response to stimulation with SARS-CoV-2 spike protein | Day 90 following initial vaccination
  Serum Sample
Quantity of TNF-a secreted in response to stimulation with SARS-CoV-2 spike protein | Day 90 following initial vaccination
  Serum Sample
Titer of antibody against SARS-CoV-2 spike protein | Day 180 following initial vaccination
  Serum Sample
Quantity of IFN-g secreted in response to stimulation with SARS-CoV-2 spike protein | Day 180 following initial vaccination
  Serum Sample
Titer of antibody against SARS-CoV-2 spike protein | 28-42 days following booster vaccination
  Serum Sample
Quantity of TNF-a secreted in response to stimulation with SARS-CoV-2 spike protein | 28-42 days following booster vaccination
  Serum Sample
Quantity of IFN-g secreted in response to stimulation with SARS-CoV-2 spike protein | 28-42 days following booster vaccination
  Serum Sample

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohan, MD PhD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Neurological Specialties West, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Study data will be kept in secure computer files, in locked research offices that are both only accessible to research personnel, and in a secure password protected Clinical Trial Management System (CTMS). Publications or presentations will report aggregate data and will not contain any subject identification.

REFERENCES:
- [Background] Kataria S, Tandon M, Melnic V, Sriwastava S. A case series and literature review of multiple sclerosis and COVID-19: Clinical characteristics, outcomes and a brief review of immunotherapies. eNeurologicalSci. 2020 Dec;21:100287. doi: 10.1016/j.ensci.2020.100287. Epub 2020 Nov 2. PMID 33163634
- [Background] Mohn N, Konen FF, Pul R, Kleinschnitz C, Pruss H, Witte T, Stangel M, Skripuletz T. Experience in Multiple Sclerosis Patients with COVID-19 and Disease-Modifying Therapies: A Review of 873 Published Cases. J Clin Med. 2020 Dec 16;9(12):4067. doi: 10.3390/jcm9124067. PMID 33339436
- [Background] Sormani MP; Italian Study Group on COVID-19 infection in multiple sclerosis. An Italian programme for COVID-19 infection in multiple sclerosis. Lancet Neurol. 2020 Jun;19(6):481-482. doi: 10.1016/S1474-4422(20)30147-2. Epub 2020 Apr 30. No abstract available. PMID 32359409
- [Background] Louapre C, Collongues N, Stankoff B, Giannesini C, Papeix C, Bensa C, Deschamps R, Creange A, Wahab A, Pelletier J, Heinzlef O, Labauge P, Guilloton L, Ahle G, Goudot M, Bigaut K, Laplaud DA, Vukusic S, Lubetzki C, De Seze J; Covisep investigators; Derouiche F, Tourbah A, Mathey G, Theaudin M, Sellal F, Dugay MH, Zephir H, Vermersch P, Durand-Dubief F, Francoise R, Androdias-Condemine G, Pique J, Codjia P, Tilikete C, Marcaud V, Lebrun-Frenay C, Cohen M, Ungureanu A, Maillart E, Beigneux Y, Roux T, Corvol JC, Bordet A, Mathieu Y, Le Breton F, Boulos DD, Gout O, Gueguen A, Moulignier A, Boudot M, Chardain A, Coulette S, Manchon E, Ayache SS, Moreau T, Garcia PY, Kumaran D, Castelnovo G, Thouvenot E, Taithe F, Poupart J, Kwiatkowski A, Defer G, Derache N, Branger P, Biotti D, Ciron J, Clerc C, Vaillant M, Magy L, Montcuquet A, Kerschen P, Coustans M, Guennoc AM, Brochet B, Ouallet JC, Ruet A, Dulau C, Wiertlewski S, Berger E, Buch D, Bourre B, Pallix-Guiot M, Maurousset A, Audoin B, Rico A, Maarouf A, Edan G, Papassin J, Videt D. Clinical Characteristics and Outcomes in Patients With Coronavirus Disease 2019 and Multiple Sclerosis. JAMA Neurol. 2020 Sep 1;77(9):1079-1088. doi: 10.1001/jamaneurol.2020.2581. PMID 32589189